CLINICAL TRIAL: NCT01464255
Title: Clinical Performance of Ocufilcon D With a Wetting Agent to Ocufilcon B
Brief Title: Comparative Study of Two Marketed 1-day Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CV-OMC-01
Record Dates: First submitted 2011-10-26; First posted 2011-11-03 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Myopia
Keywords: contact lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ocufilcon D (Experimental): Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
  Interventions: Device: ocufilcon B
- ocufilcon B (Active Comparator): Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
  Interventions: Device: ocufilcon D

INTERVENTIONS:
Device: ocufilcon D — Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
  Other Names: oculfilcon D (Daily wear soft contact lens)
  Arms: ocufilcon B
Device: ocufilcon B — Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
  Other Names: oculfilcon B (Daily wear soft contact lens)
  Arms: ocufilcon D

SUMMARY:
This study is designed to evaluate ocufilcon D lens compared to ocufilcon B lens in a 1-week crossover, daily wear regimen.

DETAILED DESCRIPTION:
This study is designed to evaluate 2 daily disposable contact lenses that are both currently cleared for the USA market. Study of the ocufilcon D lens compared to the ocufilcon B lens in a 1-week crossover, daily wear regimen. The primary objective is the comparison of fitting characteristics. The secondary objective is the comparison of comfort, end of day comfort and dryness measures.

ELIGIBILITY:
Inclusion Criteria:

* Has had a self reported oculo-visual examination in the last two years.
* Is able to wear the study lenses for at least eight hours a day, seven days a week
* Aged 18-40 years and has full legal capacity as a volunteer
* Has a distance contact lens prescription from -0.25 and -6.00D inclusive
* Has spectacle astigmatism of < 1.00D in each eye
* Baseline vision of 20/20 best-corrected in each eye.
* Is correctable to at least 20/25 distance visual acuity with study contact lenses in each eye
* Has read and understood the consent form and willing to sign consent form
* Willing and able to follow participant instructions and attend the required study visits Has worn soft contact lenses for at least two weeks prior to the study (daily wear only).

Exclusion Criteria:

* Currently wears contact lenses on an extended wear basis.
* Not a current or past wearer of the ocufilcon B 52% 1-day lenses.
* Has undergone anterior ocular surgery
* Is aphakic
* Has never worn contact lenses before
* Has any systemic disease which clinically contraindicates contact lenses
* Has active ocular disease or severe insufficiency of lacrimal secretion (dry eye)
* Use of systemic or topical medications that will affect ocular health or visual performance
* Slit lamp findings with a grading of greater than 1.0 using the grading scales in Appendix 3
* Not possible to achieve a satisfactory fit with the lens design used in the study
* Has keratoconus or other corneal irregularity
* Participating in another eye-related clinical trial
* Pregnant, lactating or planning a pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thao N Yeh, OD, Principal Investigator — U.C. Berkeley, School of Optometry
Locations (1):
- Clinical Research Center, U.C. Berkeley, School of Optometry, Berkeley, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 71 subjects were recruited for the study, with 21 subjects being disqualified at the initial screening for a total of 50 subjects started.
Pre-assignment Details: Fifty subjects started. Forty-nine subjects completed the study. One subject was disqualified after one week of wear of the control lens (ocufilcon B) during the 1st week of the study due to unresolved corneal staining.
Groups:
- Ocufilcon D Then Ocufilcon B: Participants were randomized to wear ocufilcon D lenses for 1 week and then crossed over to the ocufilcon B lens pair for 1 week.
- Ocufulcon B Then Ocufilcon D: Participants were randomized to wear ocufilcon B lenses for 1 week and then crossed over to the ocufilcon D lens pair for 1 week.
Period: Overall Study
Arm/Group | Ocufilcon D Then Ocufilcon B | Ocufulcon B Then Ocufilcon D
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — unresolve corneal staining | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 subject being disqualified after 1 week of wear
Groups:
- Ocufilcon B Then Ocufilcon D: Participants were randomized to wear ocufilcon B lenses for 1 week and then crossed over to the ocufilcon D lens pair for 1 week.
- Total: Total of all reporting groups
Arm/Group | Ocufilcon D Then Ocufilcon B | Ocufilcon B Then Ocufilcon D | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit - Decentration After Insertion
Description: The ophthalmologist's objective assessment of lens fit measurement of decentration after insertion (20 minutes settling) of Pair #1 (measured at baseline visit) and Pair #2 (measured at 7 days after baseline visit). (mm, horizontal and vertical).
Time Frame: Baseline and 7 days from baseline visit
Population: Of 49 total participants, 49 wore pair #1 and 49 crossed over to wear pair #2
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Ocufilcon D Then Ocufilcon B; Ocufilcon B Then Ocufilcon D: Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
Arm/Group | Ocufilcon D Then Ocufilcon B | Ocufilcon B Then Ocufilcon D
Number analyzed (Participants) | 49 | 49
mm
  Horizontal | 0.12 (0.29) | 0.07 (0.30)
  Vertical | -0.11 (0.47) | -0.15 (0.48)

2. Primary Outcome: Lens Fit - Decentration at One Week
Description: The ophthalmologist's objective assessment of lens fit measurement of decentration of Pair #1 (measured at 7 days after baseline visit) and Pair #2 (measured at 14 days after baseline visit). Each pair worn for one week daily disposable wear basis (at least 8 hours per day, 7 days per week). Lenses worn minimum 2 hours prior to visit. (mm, horizontal and vertical).
Time Frame: 7 days and 14 days from baseline visit
Population: Of 49 total participants, 49 wore pair #1 and 49 crossed over to wear pair #2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ocufilcon D Then Ocufilcon B | Ocufilcon B Then Ocufilcon D
Number analyzed (Participants) | 49 | 49
mm
  Horizontal | 0.14 (0.36) | 0.09 (0.37)
  Vertical | -0.08 (0.39) | -0.18 (0.51)

3. Primary Outcome: Lens Fit - Tightness After Insertion
Description: The ophthalmologist's rating of lens fit measurement of push-up tightness after insertion (20 minutes settling) of Pair #1 (measured at baseline visit) and Pair #2 (measured at 7 days after baseline visit). (0-100%, 5% steps, 0%=excessively loose, 50%=optimum, 100%=excessively tight ).
Time Frame: Baseline and 7 days from baseline visit
Population: Of 49 total participants, 49 wore pair #1 and 49 crossed over to wear pair #2
Measure: Mean (Standard Deviation); unit: percentage of tightness
Arm/Group | Ocufilcon D Then Ocufilcon B | Ocufilcon B Then Ocufilcon D
Number analyzed (Participants) | 49 | 49
percentage of tightness | 50.0 (14.1) | 52.4 (15.7)

4. Primary Outcome: Lens Fit - Tightness at One Week
Description: The ophthalmologist's rating of lens fit measurement of push-up tightness of Pair #1 (measured at 7 days after baseline visit) and Pair #2 (measured at 14 days after baseline visit). Each pair worn for one week daily disposable wear basis (at least 8 hours per day, 7 days per week). Lenses worn minimum 2 hours prior to visit. (0-100%, 5% steps, 0%=excessively loose, 50%=optimum, 100%=excessively tight ).
Time Frame: 7 days and 14 days from baseline visit
Population: Of 49 total participants, 49 wore pair #1 and 49 crossed over to wear pair #2
Measure: Mean (Standard Deviation); unit: percentage of tightness
Arm/Group | Ocufilcon D Then Ocufilcon B | Ocufilcon B Then Ocufilcon D
Number analyzed (Participants) | 49 | 49
percentage of tightness | 42.4 (12.9) | 46 (13.7)

5. Secondary Outcome: Overall Preference - Comfort After Insertion
Description: Participant's subjective rating for overall preference of lens comfort immediately after insertion for lens pair #1 or Pair #2. Surveyed at 14 days after baseline visit. (Each pair worn for one week daily disposable wear basis, at least 8 hours per day, 7 days per week). Rated by Likert scale, (forced choices - Strongly Prefer New Lenses (Week 2), Slightly Prefer New Lenses (Week 2), No Preference, Slightly Prefer Previous Lenses (Week 1), Strongly Prefer Previous Lenses (Week 1). Reported as Strongly Prefer Test Lenses, Slightly Prefer Test Lenses, No Preference, Slightly Prefer Control Lenses, Strongly Prefer Control Lenses.
Time Frame: 14 days from baseline visit
Measure: Number; unit: percentage of participants
Groups:
- Overall Study Group: Participants wore (experimental) ocufilcon D lenses or (active comparator) ocufilcon B lens bilaterally in a randomized order for 1 week and then crossed over to the alternate pair for 1 week.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 49
percentage of participants
  Strongly Prefer Test Lenses | 43
  Slightly Prefer Test Lenses | 21
  No Preference | 18
  Slightly Prefer Control Lenses | 16
  Strongly Prefer Control Lenses | 2

6. Secondary Outcome: Overall Preference - Comfort Before Removal
Description: Participant's subjective rating for overall preference of lens comfort immediately before removal for lens pair #1 or Pair #2. Surveyed at 14 days after baseline visit. (Each pair worn for one week daily disposable wear basis, at least 8 hours per day, 7 days per week). Rated by Likert scale, (forced choices - Strongly Prefer New Lenses (Week 2), Slightly Prefer New Lenses (Week 2), No Preference, Slightly Prefer Previous Lenses (Week 1), Strongly Prefer Previous Lenses (Week 1). Reported as Strongly Prefer Test Lenses, Slightly Prefer Test Lenses, No Preference, Slightly Prefer Control Lenses, Strongly Prefer Control Lenses.
Time Frame: 14 days from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 49
percentage of participants
  Strongly Prefer Test Lenses | 29
  Slightly Prefer Test Lenses | 29
  No Preference | 18
  Slightly Prefer Control Lenses | 20
  Strongly Prefer Control Lenses | 4

7. Secondary Outcome: Overall Preference - Dryness After Insertion
Description: Participant's subjective rating for overall preference of lens dryness immediately after insertion for lens pair #1 or Pair #2. Surveyed at 14 days after baseline visit. (Each pair worn for one week daily disposable wear basis, at least 8 hours per day, 7 days per week). Rated by Likert scale, (forced choices - Strongly Prefer New Lenses (Week 2), Slightly Prefer New Lenses (Week 2), No Preference, Slightly Prefer Previous Lenses (Week 1), Strongly Prefer Previous Lenses (Week 1). Reported as Strongly Prefer Test Lenses, Slightly Prefer Test Lenses, No Preference, Slightly Prefer Control Lenses, Strongly Prefer Control Lenses.
Time Frame: 14 days from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 49
percentage of participants
  Strongly Prefer Test Lenses | 23
  Slightly Prefer Test Lenses | 12
  No Preference | 55
  Slightly Prefer Control Lenses | 10
  Strongly Prefer Control Lenses | 0

8. Secondary Outcome: Overall Preference - Dryness Before Removal
Description: Participant's subjective rating for overall preference of lens dryness immediately before removal for lens pair #1 or Pair #2. Surveyed at 14 days after baseline visit. (Each pair worn for one week daily disposable wear basis, at least 8 hours per day, 7 days per week). Rated by Likert scale, (forced choices - Strongly Prefer New Lenses (Week 2), Slightly Prefer New Lenses (Week 2), No Preference, Slightly Prefer Previous Lenses (Week 1), Strongly Prefer Previous Lenses (Week 1). Reported as Strongly Prefer Test Lenses, Slightly Prefer Test Lenses, No Preference, Slightly Prefer Control Lenses, Strongly Prefer Control Lenses.
Time Frame: 14 days from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 49
percentage of participants
  Strongly Prefer Test Lenses | 33
  Slightly Prefer Test Lenses | 22
  No Preference | 25
  Slightly Prefer Control Lenses | 18
  Strongly Prefer Control Lenses | 2

9. Secondary Outcome: Overall Preference - Handling, Inserting
Description: Participant's subjective rating for overall preference of lens ease of handling at inserting for lens pair #1 or Pair #2. Surveyed at 14 days after baseline visit. (Each pair worn for one week daily disposable wear basis, at least 8 hours per day, 7 days per week). Rated by Likert scale, (forced choices - Strongly Prefer New Lenses (Week 2), Slightly Prefer New Lenses (Week 2), No Preference, Slightly Prefer Previous Lenses (Week 1), Strongly Prefer Previous Lenses (Week 1). Reported as Strongly Prefer Test Lenses, Slightly Prefer Test Lenses, No Preference, Slightly Prefer Control Lenses, Strongly Prefer Control Lenses.
Time Frame: 14 days from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 49
percentage of participants
  Strongly Prefer Test Lenses | 18
  Slightly Prefer Test Lenses | 23
  No Preference | 47
  Slightly Prefer Control Lenses | 8
  Strongly Prefer Control Lenses | 4

10. Secondary Outcome: Overall Preference - Handling, Removing
Description: Participant's subjective rating for overall preference of lens ease of handling at removing for lens pair #1 or Pair #2. Surveyed at 14 days after baseline visit. (Each pair worn for one week daily disposable wear basis, at least 8 hours per day, 7 days per week). Rated by Likert scale, (forced choices - Strongly Prefer New Lenses (Week 2), Slightly Prefer New Lenses (Week 2), No Preference, Slightly Prefer Previous Lenses (Week 1), Strongly Prefer Previous Lenses (Week 1). Reported as Strongly Prefer Test Lenses, Slightly Prefer Test Lenses, No Preference, Slightly Prefer Control Lenses, Strongly Prefer Control Lenses.
Time Frame: 14 days from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 49
percentage of participants
  Strongly Prefer Test Lenses | 8
  Slightly Prefer Test Lenses | 16
  No Preference | 74
  Slightly Prefer Control Lenses | 2
  Strongly Prefer Control Lenses | 0

11. Secondary Outcome: Overall Lens Pair Preference
Description: Participant's subjective rating for overall preference for lens pair #1 or Pair #2 based on comfort, vision and handling. Surveyed at 14 days after baseline visit. (Each pair worn for one week daily disposable wear basis, at least 8 hours per day, 7 days per week). Rated by Likert scale, (forced choices - Strongly Prefer New Lenses (Week 2), Slightly Prefer New Lenses (Week 2), No Preference, Slightly Prefer Previous Lenses (Week 1), Strongly Prefer Previous Lenses (Week 1). Reported as Strongly Prefer Test Lenses, Slightly Prefer Test Lenses, No Preference, Slightly Prefer Control Lenses, Strongly Prefer Control Lenses.
Time Frame: 14 days from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 49
percentage of participants
  Strongly Prefer Test Lenses | 43
  Slightly Prefer Test Lenses | 22
  No Preference | 2
  Slightly Prefer Control Lenses | 29
  Strongly Prefer Control Lenses | 4

12. Primary Outcome: Lens Fit - Post-Blink Lens Movement After Insertion
Description: The ophthalmologist's objective assessment of lens fit measurement of post-blink lens movement after insertion (20 minutes settling) of Pair #1 (measured at baseline visit) and Pair #2 (measured at 7 days after baseline visit). (mm).
Time Frame: Baseline and 7 days from baseline visit
Population: Of 49 total participants, 49 wore pair #1 and 49 crossed over to wear pair #2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ocufilcon D Then Ocufilcon B | Ocufilcon B Then Ocufilcon D
Number analyzed (Participants) | 49 | 49
mm | 0.29 (0.28) | 0.3 (0.32)

13. Primary Outcome: Lens Fit - Post-Blink Lens Movement Prior to Removal
Description: The ophthalmologist's objective assessment of lens fit measurement of post-blink lens movement prior to removal of Pair #1 (measured at 7 days after baseline visit) and Pair #2 (measured at 14 days after baseline visit). (mm).
Time Frame: 7 days and 14 days from baseline visit
Population: Of 49 total participants, 49 wore pair #1 and 49 crossed over to wear pair #2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ocufilcon D Then Ocufilcon B | Ocufilcon B Then Ocufilcon D
Number analyzed (Participants) | 49 | 49
mm | 0.38 (0.32) | 0.48 (0.41)

ADVERSE EVENTS:
Groups:
- Ocufilcon D; Ocufilcon B: Participants wore (experimental) ocufilcon D lenses or (active comparator) ocufilcon B lens bilaterally in a randomized order for 1 week and then crossed over to the alternate pair for 1 week.
Arm/Group | Ocufilcon D | Ocufilcon B
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor. This restriction will apply for a period of five years from completion of the study.